CLINICAL TRIAL: NCT04286659
Title: Receptor for Advanced Glycation End Products (RAGE) Polymorphisms In Inflammatory Bowel Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Noha Refaat Abdelhamid, Dr, Assiut University
Other Study IDs: Polymorphisms in IBD
Record Dates: First submitted 2020-02-25; First posted 2020-02-27 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Whole Blood Sample
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group: 90 Apparently healthy individuals
- IBD group: 90 Previously or Newly Diagnosed Ulcerative Colitis and Crohn's disease

SUMMARY:
The inflammatory bowel diseases (IBD) are chronic inflammatory disorders of the gastrointestinal tract that manifests as Crohn's disease (CD) and Ulcerative colitis (UC . Over the last two decades the incidence pattern of UC showed significant increase in previously low incidence areas such as Asia and the Middle East. In addition to microbial and environmental factors influencing IBDs, they are complex genetically, where hundreds of genetic loci contribute to disease susceptibility . Genome-wide association studies (GWAS) have identified several genetic susceptibility loci for UC and CD. Among the genetic factors involved, there are several single nucleotide polymorphisms (SNP) in molecules of the immune system associated with either susceptibility or protective effects to IBD progression, but with contradictory associations, mainly depending on the onset (adult or pediatric), sample size differences, inadequate statistical power and on the ethnicity-dependent genetic background. Growing evidence indicates that (RAGE) is involved in chronic inflammation and cancer. It is a transmembrane receptor normally expressed at low levels on a wide range of cells, bind a broad spectrum of ligands. Activated RAGE induces the synthesis of proinflammatory molecules resulting in magnifying rather than dampening inflammation . The human RAGE gene is located on chromosome 6p21.3, in the so-called class III of the major histocompatibility complex. The SNP at the -374A/T and -429T/C of the promoter region have been shown to increase protein synthesis threefold and twofold, respectively. Few studies found that RAGE is up-regulated in IBD, and it appears to play a role in the mechanisms involved in chronic inflammation Little information is available on the possible association of such polymorphisms with IBD. Few studies was carried out in different countries to assess these polymorphisms in IBD, resulting in conflicting results, between supporting and denial of the association. Due to this discrepancy we aimed to study this gene in our community including IBD patients.

DETAILED DESCRIPTION:
This study aims:

1. To investigate the association of both allelic and genotypic -374T/A and -429T/C polymorphisms and inflammatory bowel disease.
2. To correlate the relation between the studied SNPs , disease activity and the clinical features of the disease.

Subjects and Methods:

This is a case control study. The study will include 90 patients diagnosed as IBD. Patients will be recruited from outpatient department of Elraghey Liver Hospital in Assiut University Hospital.The clinical disease activity was calculated using the Montreal classification of disease activity and Crohn's Disease Activity Index (CDAI) for UC and CD patients, respectively (Silverberg et al., 2005).

-Also, 90 apparently healthy subjects (age and sex matched with the patient group) will be included as control group.

ELIGIBILITY:
Inclusion Criteria: Egyprian IBD patients Attending ElRaghy Hospital in Assuit University hopital

-

Exclusion Criteria:

* Exclusion criteria included the presence of neurological or cardiovascular diseases, diabetes, acute systemic illnesses, and previous or current history of cancer.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 90 Patients and 90 Healthy Controls
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Association Of gene polymorphisms -374T/A and -429T/C in IBD patients | 2020- 2023
  Compare the percentage of the polymorphism in Controls vs Patients

SECONDARY OUTCOMES:
To correlate the relation between the studied SNPs , disease activity and the clinical features of the disease | 2020-2023
  find If there is a relation between the Found SNPs and disease activity and feature

CONTACTS AND LOCATIONS:
Overall Officials: Elham Abdelsamie, Principal Investigator — Assiut University

REFERENCES:
- [Background] Zallot C, Peyrin-Biroulet L. Deep remission in inflammatory bowel disease: looking beyond symptoms. Curr Gastroenterol Rep. 2013 Mar;15(3):315. doi: 10.1007/s11894-013-0315-7. PMID 23354742
- [Background] Norouzinia M, Naderi N. Personalized management of IBD; is there any practical approach? Gastroenterol Hepatol Bed Bench. 2015 Winter;8(1):1-3. No abstract available. PMID 25584169
- [Background] Ng SC, Shi HY, Hamidi N, Underwood FE, Tang W, Benchimol EI, Panaccione R, Ghosh S, Wu JCY, Chan FKL, Sung JJY, Kaplan GG. Worldwide incidence and prevalence of inflammatory bowel disease in the 21st century: a systematic review of population-based studies. Lancet. 2017 Dec 23;390(10114):2769-2778. doi: 10.1016/S0140-6736(17)32448-0. Epub 2017 Oct 16. PMID 29050646
- [Background] Girardelli M, Basaldella F, Paolera SD, Vuch J, Tommasini A, Martelossi S, Crovella S, Bianco AM. Genetic profile of patients with early onset inflammatory bowel disease. Gene. 2018 Mar 1;645:18-29. doi: 10.1016/j.gene.2017.12.029. Epub 2017 Dec 15. PMID 29248579
- [Background] Sims GP, Rowe DC, Rietdijk ST, Herbst R, Coyle AJ. HMGB1 and RAGE in inflammation and cancer. Annu Rev Immunol. 2010;28:367-88. doi: 10.1146/annurev.immunol.021908.132603. PMID 20192808
- [Background] Jostins L, Ripke S, Weersma RK, Duerr RH, McGovern DP, Hui KY, Lee JC, Schumm LP, Sharma Y, Anderson CA, Essers J, Mitrovic M, Ning K, Cleynen I, Theatre E, Spain SL, Raychaudhuri S, Goyette P, Wei Z, Abraham C, Achkar JP, Ahmad T, Amininejad L, Ananthakrishnan AN, Andersen V, Andrews JM, Baidoo L, Balschun T, Bampton PA, Bitton A, Boucher G, Brand S, Buning C, Cohain A, Cichon S, D'Amato M, De Jong D, Devaney KL, Dubinsky M, Edwards C, Ellinghaus D, Ferguson LR, Franchimont D, Fransen K, Gearry R, Georges M, Gieger C, Glas J, Haritunians T, Hart A, Hawkey C, Hedl M, Hu X, Karlsen TH, Kupcinskas L, Kugathasan S, Latiano A, Laukens D, Lawrance IC, Lees CW, Louis E, Mahy G, Mansfield J, Morgan AR, Mowat C, Newman W, Palmieri O, Ponsioen CY, Potocnik U, Prescott NJ, Regueiro M, Rotter JI, Russell RK, Sanderson JD, Sans M, Satsangi J, Schreiber S, Simms LA, Sventoraityte J, Targan SR, Taylor KD, Tremelling M, Verspaget HW, De Vos M, Wijmenga C, Wilson DC, Winkelmann J, Xavier RJ, Zeissig S, Zhang B, Zhang CK, Zhao H; International IBD Genetics Consortium (IIBDGC); Silverberg MS, Annese V, Hakonarson H, Brant SR, Radford-Smith G, Mathew CG, Rioux JD, Schadt EE, Daly MJ, Franke A, Parkes M, Vermeire S, Barrett JC, Cho JH. Host-microbe interactions have shaped the genetic architecture of inflammatory bowel disease. Nature. 2012 Nov 1;491(7422):119-24. doi: 10.1038/nature11582. PMID 23128233
- [Background] Schmidt AM, Yan SD, Yan SF, Stern DM. The multiligand receptor RAGE as a progression factor amplifying immune and inflammatory responses. J Clin Invest. 2001 Oct;108(7):949-55. doi: 10.1172/JCI14002. No abstract available. PMID 11581294
- [Background] Sugaya K, Fukagawa T, Matsumoto K, Mita K, Takahashi E, Ando A, Inoko H, Ikemura T. Three genes in the human MHC class III region near the junction with the class II: gene for receptor of advanced glycosylation end products, PBX2 homeobox gene and a notch homolog, human counterpart of mouse mammary tumor gene int-3. Genomics. 1994 Sep 15;23(2):408-19. doi: 10.1006/geno.1994.1517. PMID 7835890
- [Background] Hudson BI, Stickland MH, Futers TS, Grant PJ. Effects of novel polymorphisms in the RAGE gene on transcriptional regulation and their association with diabetic retinopathy. Diabetes. 2001 Jun;50(6):1505-11. doi: 10.2337/diabetes.50.6.1505. PMID 11375354
- [Background] Ciccocioppo R, Bozzini S, Betti E, Imbesi V, Klersy C, Lakyova LS, Sukovsky L, Benacka J, Kruzliak P, Corazza GR, Di Sabatino A, Falcone C. Functional polymorphisms of the receptor for the advanced glycation end product promoter gene in inflammatory bowel disease: a case-control study. Clin Exp Med. 2019 Aug;19(3):367-375. doi: 10.1007/s10238-019-00562-x. Epub 2019 Jun 7. PMID 31175506